CLINICAL TRIAL: NCT06855654
Title: Promoting Resilience in Stress Management for Metastatic Breast Cancer (PRISM-MBC)
Brief Title: Promoting Resilience in Women With Breast Cancer (PRISM -MBC)
Acronym: PRISMMBC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LCCC2424
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Metastatic Breast Cancer
Keywords: Promoting Resilience in Women with Breast Cancer (PRISM); remote; Black women; adverse social determinants of health
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRISM (Experimental): Participants with metastatic breast cancer (MBC) receive the Promoting Resilience in Women with Breast Cancer (PRISM) intervention.
  Interventions: Behavioral: Promoting Resilience in Women with Breast Cancer (PRISM)

INTERVENTIONS:
Behavioral: Promoting Resilience in Women with Breast Cancer (PRISM) — PRISM is a brief, skills-based intervention targeting 4 core resilience resources (stress management, goal setting, cognitive reframing, and meaning-making) followed by an optional family session. This adapted version of the PRISM intervention will be delivered1:1 by trained coaches who speak English or Spanish via HIPAA-compliant video conference.A single coach conducts the program with a single patient. Each session is 30-60 minutes, for a total of 2- 4 hours. Sessions are delivered every 1-2 weeks per patient's preference. To facilitate on-demand skills-practice between sessions, all participants have access to the PRISM app, available for iOS/Android, and thus available to the >90% of U.S. adults who own a smartphone. Participants will be assisted to download the PRISM app to their device at the time of registration; however, coaches can also provide assistance with app access during intervention sessions.

SUMMARY:
This pilot interventional study evaluates the change from baseline to post-intervention in resilience and other patient-reported outcomes for individuals with a recent diagnosis of metastatic breast cancer (MBC) participating in the Promoting Resilience in Women with Breast Cancer (PRISM) intervention, overall and stratified by race, and to evaluate the feasibility and acceptability of the PRISM intervention in the MBC population.

Black women with MBC have shorter survival from the time of metastatic diagnosis to death, compared to White women with clinically similar disease, and may have more rapid declines in quality of life over time. Adverse social determinants of health may play a role in these outcome disparities, due to both social barriers in accessing care, and through direct stress-mediated biological effects on the host and tumor microenvironment. Interventions to reduce stress and optimize resilience during treatment of MBC may improve quality of life and even improve disease outcomes; however, feasibility of face-to-face intervention during intensive medical treatment is limited. Thus, this study aims to demonstrate the feasibility of a remotely delivered resilience intervention, PRISM, already proven effective in other cancer settings, for MBC patients, and to gather preliminary efficacy data for a future randomized trial.

DETAILED DESCRIPTION:
Black women with breast cancer have substantially worse survival compared to White counterparts across all stages of presenting disease. Survival from a diagnosis of metastatic breast cancer (MBC) to death is shorter for Black compared to non-Black women, with the worst disparity appearing in younger patients.

Black compared to non-Black MBC patients also report more chronic stressors including social barriers to cancer care, metabolic co-morbidities, and higher likelihood of residing in neighborhoods with adverse social determinants of health (SDOH). These bio-psycho-social factors are potential mechanisms of observed racial gaps in survival of MBC. The adversity experienced by Black patients may impact the outcomes of MBC through social, psychological, and biological mechanisms. Regarding social mechanisms, adverse SDOH may cause patients to have delays in care, miss appointments, defer needed treatment, or tolerate treatment less well due to unmet supportive care or social support needs. Regarding psychological and biological mechanisms, cumulative physiologic stress and distress elevate inflammatory and immune biomarkers and precipitate the development of cardio-metabolic diseases, a phenomenon known as allostatic overload. Black individuals both with and without cancer are more likely to suffer from allostatic overload, and the impact of cancer on allostatic load may be differential by race. While the Black-White gap in breast cancer survival has long been recognized, the relationships among marginalized racial identity, adverse social circumstances, allostatic overload, and breast cancer outcomes remain poorly understood.

Stress and Coping Theory posits that the ways in which individuals appraise and cope with stressful experiences are modifiable targets for intervention. In this regard, "resilience" is a key construct; it implies an ability to harness resources to sustain well-being in the face of adversity. In breast cancer patients and others with serious illness, skills in stress-management, goal-setting, positive-reframing, and meaning - making are associated with improved stress biology, physical, and mental health. In the context of an advanced cancer diagnosis, resilient individuals may be more able to cope with the challenges of illness, including barriers to care, and in turn experience less incremental stress, and improved quality of life (QOL) and disease outcomes. Such resilience might be particularly beneficial to patients from marginalized groups.

Investigators of this study have previously developed and demonstrated the efficacy of a targeted intervention promoting resilience in populations of young adults with pediatric cancers and advanced cancers. However, evidence is lacking as to whether such an intervention can be helpful among women with MBC, particularly those from historically marginalized communities. The goal of this study is to test the impacts of a remotely delivered resilience intervention, Promoting Resilience in Stress Management (PRISM), on relevant social, psychological, and biologic outcomes of diverse women with a recent diagnosis of MBC at the University of North Carolina-Chapel Hill (UNC) and the University of Alabama-Birmingham (UAB).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained to participate in the study and HIPAA authorization for release of personal health information.
* Participants are willing and able to comply with study procedures based on the judgement of the investigator.
* Male and female patients of age >18 years.
* Pathologic diagnosis of metastatic breast cancer within 182 days prior to enrollment date.
* Able to answer surveys and participate in counseling sessions in English (the patient's first language is not required to be English).
* Indicate intent to receive ongoing cancer care at the enrolling institution.

Exclusion Criteria:

Individuals meeting any of the following exclusion criteria will be excluded from study participation.

* Patient unwilling or unable to complete surveys via one of the following methods: (a) paper survey completed in clinic or mailed directly to patient's home address, including a pre-addressed, pre-stamped return envelope in the mailed survey packet, or (b) electronic survey links sent via emails or text link on a mobile device, tablet, laptop, or desktop computer.
* Patient unwilling or unable to provide verbal or signed consent to participate.
* Participant cannot read English.
* Patient has permanently discontinued cancer-directed therapy or does not intend to receive any cancer-directed therapy, is receiving home or residential hospice care, is hospitalized, or is described as likely to die within 90 days or actively dying in last provider documentation, at the time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Resilience Score Change | Baseline and 3 months
  Resilience Score Change will be assessed baseline to 3 months using Connor Davidson Resilience Score, overall and stratified by race (Black/non-Black).

SECONDARY OUTCOMES:
Change in allostatic load index (ALI) | Baseline and 12 months
  Change in allostatic load index (ALI) including glycosylated Hgb, total cholesterol, HDL, LDL, triglycerides, high-sensitivity C-reactive protein, albumin and creatinine from pre- to post-intervention, overall, and stratified by race (Black/non-Black) will be reported.
Time to progression | Baseline and 12 months
  Time to progression is the length of time from baseline until the disease begins to spread or worsen will be reported among PRISM participants, stratified by race.
Survival | Baseline and 12 months
  Survival is defined as the time from baseline to date of death for any cause will be reported among PRISM participants, stratified by race.

CONTACTS AND LOCATIONS:
Overall Officials: Katie Reeder-Hayes, MD, MBA, MSCR, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (2):
- United States (2):
  - The University of Alabama, Birmingham, Alabama
  - University of North Carolina, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical trials at UNC Lineberger — http://unclineberger.org/patientcare/clinical-trials/clinical-trials